CLINICAL TRIAL: NCT07092306
Title: A Randomized Controlled Study Comparing the Safety and Efficacy of Irinotecan Hydrochloride Liposome Injection Combined With Temozolomide and Vincristine (NALIRI-VT) Versus Irinotecan Combined With Temozolomide and Vincristine (VIT) in Patients With Advanced Ewing's Sarcoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tang Xiaodong (Other)
Responsible Party: Sponsor-Investigator, Tang Xiaodong, professor, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025PHD002-001
Record Dates: First submitted 2025-06-29; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Ewing's Sarcoma
Keywords: Irinotecan Hydrochloride Liposome Injection; NALIRI-VT; Temozolomide; Vincristine; Ewing's Sarcoma
MeSH Terms: conditions — Sarcoma, Ewing | interventions — Temozolomide; Vincristine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irinotecan Hydrochloride Liposome Injection Combined with Temozolomide and Vincristine (NALIRI-VT) (Experimental)
  Interventions: Drug: Irinotecan Hydrochloride Liposome Injection Combined with Temozolomide and Vincristine (NALIRI-VT)
- Irinotecan Combined with Temozolomide and Vincristine (VIT) (Active Comparator)
  Interventions: Drug: Irinotecan Combined with Temozolomide and Vincristine (VIT)

INTERVENTIONS:
Drug: Irinotecan Hydrochloride Liposome Injection Combined with Temozolomide and Vincristine (NALIRI-VT) — （NALIRI-VT，Nanoliposomal Irinotecan，Vincristine，Temozolomide）， Nanoliposomal Irinotecan：35 mg/m2/d，iv，D1，8，15， Temozolomide：100 mg/m2/d，po，D1-5， Vincristine：1.4 mg/m2/d，iv，D1，最大剂量2mg；
  Arms: Irinotecan Hydrochloride Liposome Injection Combined with Temozolomide and Vincristine (NALIRI-VT)
Drug: Irinotecan Combined with Temozolomide and Vincristine (VIT) — （VIT，Vincristine，Irinotecan，Temozolomide） Irinotecan：50 mg/m2/d，iv，D1-5， Temozolomide：100 mg/m2/d，po，D1-5， Vincristine：1.4 mg/m2/d，iv，D1，最大剂量2mg；
  Arms: Irinotecan Combined with Temozolomide and Vincristine (VIT)

SUMMARY:
This study is a randomized, controlled, multicenter, prospective clinical trial with a planned enrollment of 74 patients, who will be randomly assigned in a 2:1 ratio. After enrollment, patients will receive either irinotecan liposomal injection combined with temozolomide and vincristine or irinotecan injection combined with temozolomide and vincristine. The aim is to evaluate the efficacy, safety, and impact on quality of life of the irinotecan liposomal combination regimen compared to the irinotecan injection combined with temozolomide and vincristine in the treatment of advanced Ewing's sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* 1. The subject or their legal representative must sign the written informed consent before enrollment.

  2. Age ≥ 8 years and ≤ 40 years, both male and female are eligible. 3. Pathologically confirmed Ewing's sarcoma, and detailed pathological reports must be provided. Pathology must be confirmed by fluorescence in situ hybridization (FISH) or next-generation sequencing (NGS) to show the presence of Ewing's sarcoma-specific FET family (including EWSR1 or FUS) gene breaks. This study does not impose special restrictions on fusion partner genes, but clear FET-non ETS fusions (such as EWSR1-WT1, EWSR1-NFATC2, EWSR1-PATZ1, etc.) do not meet the enrollment criteria.

  4. At least one measurable target lesion as judged by RECIST 1.1 criteria. 5. Failure of first-line standard treatment. First-line standard treatment includes the following drugs: doxorubicin, cyclophosphamide and/or ifosfamide. Treatment failure is defined as disease progression during adjuvant chemotherapy or within 6 months after chemotherapy. For disease progression more than 6 months after chemotherapy, the consent of the subject or their legal representative is required.

  6. ECOG score: 0-1. 7. Expected survival ≥ 3 months. 8. Recovery from previous treatment: According to NCI-CTCAE 5.0, all side effects (except alopecia) must have subsided to grade 1 or below.

  9. Normal major organ function, meeting the following criteria:

  1) Blood routine examination must meet the following criteria (no blood transfusion, no use of hematopoietic factors, and no drug correction within 14 days):
  1. ANC ≥ 1.5×109/L;
  2. HB ≥ 90 g/L;
  3. PLT ≥ 100×109/L; 2) Biochemical examination must meet the following criteria:

  <!-- -->

  1. TBIL ≤ 1.5 ULN;
  2. ALT, AST ≤ 2.5 ULN (if liver function abnormalities are due to liver metastasis, then ≤ 5 ULN);
  3. Serum creatinine sCr ≤ 1.5 ULN, endogenous creatinine clearance rate ≥ 50 ml/min (Cockcroft-Gault formula); 3) Coagulation function must meet the following criteria: INR ≤ 1.5 and APTT ≤ 1.5 ULN.

     10. Women of childbearing age must have taken reliable contraceptive measures or undergone a pregnancy test (serum or urine) within one week before enrollment, with a negative result, and be willing to use appropriate contraceptive methods during the trial and for 8 weeks after the last administration of the investigational drug. For men, they must agree to use appropriate contraceptive methods during the trial and for 8 weeks after the last administration of the investigational drug or have undergone surgical sterilization.

     Exclusion Criteria:
* 1. Known hypersensitivity, anaphylaxis or intolerance to irinotecan liposome, temozolomide and vincristine or their excipients; 2. Within 2 weeks after the last systemic cytotoxic drug treatment, radiotherapy, targeted therapy or any anti-tumor drug treatment except immunotherapy; 3. Patients who have received irinotecan treatment before; 4. Other malignant tumors within the past 5 years; 5. Known symptomatic central nervous system metastases; 6. Known symptomatic brain metastases, spinal cord compression, carcinomatous meningitis, or unstable brain or leptomeningeal disease found on CT or MRI at screening; 7. Symptomatic serous cavity effusion (including pleural effusion, ascites, pericardial effusion) requiring surgical intervention; 8. Uncontrolled concomitant diseases, including but not limited to: poorly controlled hypertension, heart failure, diabetes, persistent active infection, poorly controlled active peptic ulcer, or mental disorders or social conditions that may affect the subject's compliance with the study; 9. Abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN + 4s or APTT > 1.5 ULN), with bleeding tendency or receiving thrombolytic or anticoagulant therapy; 10. Treatment with anticoagulants or vitamin K antagonists such as warfarin, heparin or similar drugs; Note: Under the condition of INR ≤ 1.5, low-dose heparin (adult daily dose of 6,000 - 12,000 U), low-dose aspirin (daily dose ≤ 100 mg), or rivaroxaban (daily dose ≤ 10 mg) for preventive purposes is allowed; 12. History of drug abuse of psychotropic drugs and unable to quit or with mental disorders; 13. Known hereditary or acquired bleeding and thrombotic tendencies (such as hemophilia, coagulation disorders, thrombocytopenia, hypersplenism, etc.); 14. Open wounds, fractures, or poorly healing wounds; 15. Major surgery within 2 weeks; 16. Confirmed inflammatory bowel disease, intestinal obstruction or chronic diarrhea; 17. Cavity organ fistula or perforation within 6 months; 18. Active hepatitis B or C virus infection or active infection requiring antimicrobial treatment (such as the use of antibacterial drugs, antiviral drugs, antifungal drugs); 19. Participation in other interventional anti-tumor clinical trials within 4 weeks; 20. Patients who have used strong CYP3A4 inducers or strong CYP3A4 inhibitors or strong UGT1A1 inhibitors within 3 weeks before the first dose; 21. Lactation; 22. Any condition that the investigator deems may harm the patient or prevent the patient from meeting or fulfilling the study requirements.

Ages: 8 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate，ORR | 6 weeks

SECONDARY OUTCOMES:
progression free survival，PFS | 1 year
overall survival，OS | 1 year

IPD SHARING:
Plan to Share IPD: Yes